CLINICAL TRIAL: NCT04065958
Title: Yoga-mindfulness for Pain Management in Inflammatory Arthritis - a Pragmatic Randomized Controlled Trial
Brief Title: Yoga-mindfulness for Pain Management in Inflammatory Arthritis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: 1st: Covid-19 pandemic. 2nd: Lack of resources
Sponsor: Karolinska Institutet (Other)
Collaborators: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Jon Lampa, MD, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-88
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Pain
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Pain | interventions — Patient Education as Topic; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga-mindfulness (Experimental): Yoga-mindfulness program consisting of movements/postures (asanas), breathing practices, relaxation practices and meditation practices, together with brief talks on yoga-based coping strategies. The intervention starts with a introductory lecture and is then followed by one session per week, á 90 minutes, for 15 weeks, with home assignments for about 30 minutes per day, four days per week.
  Interventions: Behavioral: Yoga-mindfulness
- Patient education and physiotherapy (Active Comparator): Patient education program consisting of lectures on topics related to inflammatory arthritis and pain together with mild physiotherapy. The interventions starts with an introductory lecture and is then followed by one session per week, á 90 minutes, for 15 weeks. Each session consists of a lecture and a program of instructed physiotherapy. Besides the weekly sessions, home assignments consisting of 30 minutes of walking, are performed four days per week.
  Interventions: Behavioral: Patient education and physiotherapy

INTERVENTIONS:
Behavioral: Yoga-mindfulness — Body-mind therapy
  Arms: Yoga-mindfulness
Behavioral: Patient education and physiotherapy — Lectures and physiotherapy
  Arms: Patient education and physiotherapy

SUMMARY:
This study evaluates the potential effects on pain, pain-related symptoms and quality of life of a yoga-mindfulness program, compared to patient education and physiotherapy, for patients with inflammatory arthritis and persistent pain problems.

DETAILED DESCRIPTION:
Earlier studies has indicated that body-mind therapies such as yoga and tai chi might be beneficial in the management of chronic pain syndromes. Chronic pain affects a large number of patients with inflammatory arthritis. Effective treatments are lacking for this patient group, so new treatment strategies are warranted.

The study is designed as randomized controlled trial where participants are allocated on a 1:1 ratio to either a 15 week intervention program of yoga-mindfulness or 15 weeks of patient education and mild physiotherapy.

Study outcomes include pain levels and other pain-related features such as fatigue, sleep problems, mood disturbances and functional disability as well as measurements of health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject has a diagnosis of either rheumatoid arthritis or psoriatic arthritis
* Subject has a total score on SIQR above 33
* Subject has not changed anti-rheumatic or analgetic treatment strategies during the three months preceding study inclusion (dose changes of ongoing treatments are accepted)

Exclusion Criteria:

* Subject has another medical condition that might prevent the subjects full participation in the interventions
* Subject has more than four swollen joints
* Subject has a C-Reactive Protein more than 20 mg/L
* Subject is currently practicing yoga or has practiced yoga regularly during the last six months prior to study inclusion
* Subject does not speak Swedish
* Subject is unwilling to comply with the study protocol
* Subject is considered, by the investigator, to be an unsuitable candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Symptom Impact Questionnaire- Revised (SIQR) | At baseline, after 5, 10 and 15 weeks of intervention as well as 12 weeks after the intervention period.
  SIQR is a questionnaire that captures the spectrum of symptoms usually associated to fibromyalgia. It consists of three domains (function, overall impact and symptoms) and includes questions about functional disability, level of disease burden and symptoms such as pain and pain-related features, e.g. fatigue, sleep problems, depression/anxiety etc. It is calculated into a score ranging from 0-100, where 0 means no symptoms. The score will be evaluated as change from baseline to study completion.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) | At baseline, after 5, 10 and 15 weeks of intervention as well as 12 weeks after the intervention period.
  Overall impression of change in symptoms during the study period. PGIC consists of a 7-point scale, ranging from 1 (Very Much Improved) to 7 (Very Much Worse).
Chronic Pain Acceptance Questionnaire (CPAQ) | At baseline, after 5, 10 and 15 weeks of intervention as well as 12 weeks after the intervention period.
  Nineteen items form the CPAQ (Wicksell et al. Eur J Pain. 2009;13(7):760-8) assessing coping strategies and acceptance in relation to chronic pain. The 19 items are divided in two categories: Activity engagement and Pain willingness. The items are rated on a 7-point scale from 0 (never true) to 6 (always true). For Activity engagement the scores are summed and for Pain willingness the scores are reversed and then summed. To obtain the total score, the scores for each category are summed. The total score ranges from 0-114, with higher scores indicating higher level of acceptance.
Pain Catastrophizing Scale (PCS) | At baseline, after 5, 10 and 15 weeks of intervention as well as 12 weeks after the intervention period.
  Assessment of negative thoughts ("catastrophizing") in relation to pain. PCS is a 13-item instrument, where each item is rated on a 5-point scale ranging from 0 (not at all) to 4 (all the time). The PCS yields a total score and three subscale scores assessing rumination, magnification and helplessness. The PCS total score is computed by summing responses to all 13 items. Total score ranges from 0-52, where a higher number indicates more catastrophizing. The rumination subscale ranges from 0-16, the magnification subscale ranges from 0-12 and the helplessness subscale ranges from 0-24.
Karolinska Sleep Questionnaire - 7 items (KSQ) | At baseline, after 5, 10 and 15 weeks of intervention as well as 12 weeks after the intervention period.
  Seven questions from the KSQ, assessing of features of sleep quality. Each questions is scored on 6 levels, from 0-5. The scores are summed to produce a global score (range 0-35). Higher scores indicate worse sleep quality.
Short Form-36 (SF-36) | At baseline, after 5, 10 and 15 weeks of intervention as well as 12 weeks after the intervention period.
  Assessment of health-related quality of life (HRQoL). SF-36 evaluates HRQoL in eight components, each component is scored on a scale ranging from 0-100, where higher scores indicate a more favorable health state.
Individual domains of SIQR | At baseline, after 5, 10 and 15 weeks of intervention as well as 12 weeks after the intervention period.
  Each of the three domains of SIQR will be assessed separately. The "function" domain ranges from 0-30, with higher scores indicating more functional disability. The "overall impact" domain ranges from 0-20 with higher scores indicating a larger overall impact. The "symptom" domain ranges from 0-50 with higher scores indicating more symptoms.
Visual Analog Scale (VAS) of pain, fatigue and general health | At baseline, after 5, 10 and 15 weeks of intervention as well as 12 weeks after the intervention period.
  Commonly assessed features in inflammatory arthritis, depicted on VAS-scales. The scales range from 0-100, with higher scores indicating worse symptoms.
Pain distribution | At baseline, after 5, 10 and 15 weeks of intervention as well as 12 weeks after the intervention period.
  Pain distribution, depicted on a pain mannequin.
Disease Activity Score, 28 joints (DAS28) | At baseline and after 15 weeks of intervention.
  Disease activity measure used in rheumatic joint diseases. Constitutes a composite score based on an assessment of number of swollen and tender joints as well as inflammatory markers in blood samples and both patients and physicians ratings of disease activity. The score ranges from 0-9.4 with higher scores indicating worse symptoms.
Hospital Anxiety and Depression Scale (HADS) | At baseline, after 5, 10 and 15 weeks of intervention as well as 12 weeks after the intervention period.
  HADS contains 14 items assessing features of anxiety and depression. Each question is scored on a 4-level scale (ranging from 0-3). Seven of the questions assess features of anxiety and the other seven questions assess features of depression. Each subscale has a total range of 0-21 with higher scores indicating worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Lampa, MD, As.Prof., Principal Investigator — Karolinska University Hospital / Karolinska Institute
Locations (2):
- Sweden (2):
  - University Hospital Örebro, Örebro
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang C, Schmid CH, Rones R, Kalish R, Yinh J, Goldenberg DL, Lee Y, McAlindon T. A randomized trial of tai chi for fibromyalgia. N Engl J Med. 2010 Aug 19;363(8):743-54. doi: 10.1056/NEJMoa0912611. PMID 20818876
- [Result] Carson JW, Carson KM, Jones KD, Bennett RM, Wright CL, Mist SD. A pilot randomized controlled trial of the Yoga of Awareness program in the management of fibromyalgia. Pain. 2010 Nov;151(2):530-539. doi: 10.1016/j.pain.2010.08.020. PMID 20946990